CLINICAL TRIAL: NCT00776542
Title: Single Dose Two-Way Crossover Fasted Bioequivalence Study of Minocycline 100 mg Capsules in Healthy Volunteers
Brief Title: Bioequivalence Study of Minocycline 100mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AAI-US-134
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence Minocycline Tablets
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Minocycline 100 mg tablets of ranbaxy
  Interventions: Drug: Minocycline 100mg Tablets
- 2 (Active Comparator): Minocin 100mg tablets
  Interventions: Drug: Minocycline 100mg Tablets

INTERVENTIONS:
Drug: Minocycline 100mg Tablets

SUMMARY:
The purpose of this study was to determine the bioequivalence of Minocycline formulations after administration of single doses to normal healthy subjects under fasted conditions. These data were to be evaluated statistically to determine if the products meet bioequivalence criteria.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover , bioequivalence study on minocycline comparing minocycline 100mg tablets of Ranbaxy pharmaceuticals inc with Minocin 100mg capsules of in healthy, adult, human, subjects under fasting conditions.

A total of 28 non-smoking subjects (16 men and 12 women) were included in this study, of which 28 finished the study according to the protocol,

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between 18 and 45 years of age inclusive.
* Informed o'f the nature of the study and given written informed consent.
* Have a body weight within 15 % of the appropriate range as defined in the 1983 Metropolitan Life Company tables and weighing at least 100 lbs.

Exclusion Criteria:

* Hypersensitivity to Minocycline (Minocin®), or other antibiotics.
* Any history of a clinical condition which might affect drug absorption, metabolism or excretion.
* Recent history of mental illness, drug addiction, drug abuse or alcoholism.
* Donation of greater than 500 ml of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.
* Received an investigational drug within the 4 weeks prior to study dosing.
* Currently taking any prescription medication, except oral contraceptives, within the 7 days pr/or to study dosing or over-the-counter medication within 3 days of study dosing. This prohibitor~ does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physic/an2
* Tobacco use (>5 cigarettes per day) in the 3 months prior to study dosing.
* If female, the subject is lactating or has a positive pregnancy test at screening and prior to each of the two treatment periods.
* Females of child bearing potential must use a 'medically acceptable method of contraception throughout the entire study period and for one week after the study is completed.
* Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral contraceptives, progestin injection' or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization of their partner(s) or abstinence.
* Females taking oral contraceptives must have taken them consistently for at least three months prior to receiving study medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2002-10; Primary Completion 2002-11 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- AII pharma, Chapell Hill, North Carolina, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html